CLINICAL TRIAL: NCT05068973
Title: Evaluation of the Performance and Tolerance of the NOVATECH ® LUCIOLA TM EB Fiducial Marker During Radiotherapy Sessions in Patients Suffering From Lung Cancer: Multicenter, Post CE-mark Study
Brief Title: Evaluation of the NOVATECH ® LUCIOLA TM EB Fiducial Marker During Radiotherapy Sessions in Lung Cancer Patients
Acronym: LUCIOLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Collaborators: NOVATECH SA (Unknown)
Responsible Party: Principal Investigator, ESCARGUEL Bruno, Pulmonologist, Hospital St. Joseph, Marseille, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LUCIOLA 2020_10_02
Record Dates: First submitted 2021-09-20; First posted 2021-10-06 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer
Keywords: Fiducial marker; Bronchoscopy; SBRT; Radiotherapy; NOVATECH LUCIOLA EB
MeSH Terms: conditions — Lung Neoplasms | interventions — Fiducial Markers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luciola (Experimental): Bronchoscopic implantation of the fiducial marker NOVATECH® LUCIOLA™ EB prior to radiotherapy treatment.
  Interventions: Device: NOVATECH® LUCIOLA™ EB - (Fiducial Marker)

INTERVENTIONS:
Device: NOVATECH® LUCIOLA™ EB - (Fiducial Marker) — Bronchoscopic implantation in the lung of the NOVATECH® LUCIOLA™ EB fiducial marker

SUMMARY:
Following CE certification, this Post Market Clinical Follow-up investigates the performance and safety of using the new fiducial marker, NOVATECH® LUCIOLA™ EB, in the lung airways to monitor in real-time tumor location during radiotherapy.

At the time of insertion near the tumor, the Luciola's 3 fiducial marker arms are deployed simultaneously. Optimal detection of the fiducial marker is considered during the radiotherapy treatment.

DETAILED DESCRIPTION:
NOVATECH® LUCIOLA™ EB fiducial marker will be implanted near the lung tumor by bronchial endoscopy by a pulmonologist. Following a dosimetry visit, participants will be proposed a maximum of 5 radiation therapy sessions. A follow-up visit at 3 months will take place after the last radiotherapy session. The participation period for each participant will be between 4.5 and 6 months. This study will evaluate the Luciola implant's performance and safety (visibility, migration, complications, tumoral response).

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years of age
* Participants with primary, secondary or metastatic lung cancer with an indication for radiotherapy and placement of a fiducial marker
* Participants who will be able to tolerate the flexible bronchoscopic implantation procedure and radiotherapy treatment.
* Participants who give their written informed consent

Exclusion Criteria:

* Participants with uncontrolled infection / participants with active infections.
* Participants with a bronchoscopy contra-indication
* Pregnant or breast-feeding women
* Participants with known allergy to one of the components (tantalum and nickel titanium alloy for the marker and polymer materials which are contained in the delivery device)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
LUCIOLA implant's performance during radiotherapy (RT) treatment: tracking rate | Takes place 4-6 weeks after implantation
  Number of RT sessions during which the LUCIOLA implant was used for treatment in relation to the total number of RT sessions.
  If LUCIOLA can be detected and used for treatment, the patient will attend 3 to 5 RT sessions over a period lasting 1 to 2 weeks.

SECONDARY OUTCOMES:
Luciola implant "visibility" | From the dosimetry visit (week 2-4 after implantation) to the last RT session (3-4 weeks after dosimetry)
  Average of the visibility rate (number of visible LUCIOLA implant arm(s) (0,1,2 or 3) compared to the total number of LUCIOLA implant arms (3)) for all the LUCIOLA implants for the entire radiotherapy treatment
Global migration rate | Dosimetry CT-Scan takes place 2-4 weeks after implantation; End of treatment CT-Scan takes place 12 weeks after last radiotherapy session
  Number of LUCIOLA implants which have migrated between the beginning (dosimetry visit) and end of treatment follow-up (12 weeks after last radiotherapy session) in relation to the total number of LUCIOLA implants
Adverse events | 4.5 to 6 months (from implantation to the end of participant's enrollment in the study)
  Occurrence rate of adverse or unexpected events which took place between implantation and up to 3 months following the RT treatment's end.
Replanning radiotherapy treatment | During radiotherapy sessions (4-6 weeks after implantation)
  Replanning rate = Number of replanning versus total number of sessions for all of the participants.
Radiotherapist's satisfaction | End of study visit: 12 weeks after last radiotherapy session
  Number of participants for whom the radiotherapist is "satisfied" in relation to the total number of participants.
Pulmonologist's satisfaction | Within 24 hours after implantation
  Number of procedures at the end of which the pulmonologist is "satisfied" in relation to the total number of procedures
  The following questions will be considered:
  * Easy introduction of the LUCIOLA delivery system in the guide sheath
  * Easy placement (release) of the LUCIOLA device at the implantation site
  * Change of the position after LUCIOLA implant release
Tumoral response | Between the inclusion CT-Scan (8 weeks prior to implantation at the most) and the radiotherapy end of treatment CT-Scan (12 weeks after last RT session)
  Tumoral response rate according to RECIST criteria between the inclusion CT-Scan and the radiotherapy end of treatment CT-Scan.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Escarguel, MD, Principal Investigator — Hôpital Saint Joseph, Marseille France
Locations (5):
- France (5):
  - Centre de radiothérapie Francois Baclesse, Caen
  - Hopital Saint Joseph, Marseille
  - Hôpital Privé Clairval-Ramsay Santé, Marseille
  - CHU Rouen, Rouen
  - Centre de radiothérapie Henri Becquerel, Rouen